CLINICAL TRIAL: NCT03343795
Title: Oral Versus Parental Progesterone in the Management of Preterm Labor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPTL
Record Dates: First submitted 2017-11-11; First posted 2017-11-17 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group 1 (Experimental): oral progesterone
  Interventions: Drug: oral progesterone
- study group 2 (Active Comparator): intramuscular progesterone
  Interventions: Drug: intramuscular progesterone

INTERVENTIONS:
Drug: oral progesterone — daily
  Arms: study group 1
Drug: intramuscular progesterone — every week
  Arms: study group 2

SUMMARY:
Preterm birth, defined as delivery at less than 37 weeks gestation, complicates approximately 12% of pregnancies in the United States

Preterm delivery has been, and remains, the most important challenge to modern obstetrics. In 2009, 13 million babies were born preterm, 11 million in Africa and Asia and 500,000 in the USA, The highest rates of preterm birth are in Africa (11.9%) and North America (10.6%)

ELIGIBILITY:
Inclusion Criteria:

1. Past history of one or more spontaneous preterm labor.
2. Singleton pregnancy.
3. Pregnancy of less than 20 weeks of gestation

Exclusion Criteria:

1. Women on tocolytic drugs .
2. Underwent cervical cerclage in this pregnancy .
3. Multiple gestations .
4. Major fetal congenital malformations .
5. Pregnancy 0f more than 20 weeks gestation .

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2018-05-13 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
the rate of preterm labor | 10 weeks
  number of women delivered before 37 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt